CLINICAL TRIAL: NCT03236961
Title: Optimizing the Antibiotic Treatment of Uncomplicated Acute Appendicitis: a Prospective Randomised Multicenter Study (The APPAC II Study)
Brief Title: Optimizing the Antibiotic Treatment of Uncomplicated Acute Appendicitis
Acronym: APPACII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other); Mikkeli Central Hospital (Other); Lapland Central Hospital (Unknown); Jyväskylä Central Hospital (Other); Satakunta Central Hospital (Other); Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, MD, PhD, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPAC II
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Acute Appendicitis
Keywords: uncomplicated acute appendicitis; complicated acute appendicitis; antibiotic therapy
MeSH Terms: conditions — Appendicitis | interventions — Ertapenem; Levofloxacin; Metronidazole; Moxifloxacin

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous & per oral antibiotics (Active Comparator): Ertapenem 1 g x 1 for two days i.v. followed by p.o. levofloxacin 500 mg x 1 and metronidazole 500 mg x 3 for 5 days, duration of treatment one week.
  Interventions: Drug: Ertapenem
- Per oral antibiotics (Active Comparator): Moxifloxacin 400 mg x 1 foe seven days, duration of treatment one week.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Ertapenem — I.v. ertapenem 1 g for 2 days followed by p.o. levofloxacin 500 mg x1 and metronidazole 500 mg x 3 for 5 days
  Other Names: Levofloxacin; Metronidazole
  Arms: Intravenous & per oral antibiotics
Drug: Moxifloxacin — P.o. moxifloxacin 400 mg x1 for 7 days
  Arms: Per oral antibiotics

SUMMARY:
Appendicectomy has been the treatment of acute appendicitis for over a hundred years. Appendicectomy, however, includes operative and postoperative risks despite being a routine procedure. Several studies have proved promising results of the safety and efficiency of antibiotics in the treatment of acute uncomplicated appendicitis. The APPAC study by the investigators, published in 2015 in the Journal of American Medical Association, also proved promising results with 73% of patients with uncomplicated appendicitis treated successfully with antibiotics. None of the patients initially treated with antibiotics that later had appendectomy had major complications. The results of the APPAC trial suggest that CT proven uncomplicated acute appendicitis is not a surgical emergency and antibiotic therapy is a safe first-line treatment option. Reducing unnecessary appendectomies has also been shown to lead to significant economic savings.

The aim of this randomized prospective study is to optimize antibiotic therapy for uncomplicated acute appendicitis by comparing different antibiotic regimens; intravenous antibiotic (ertapenem) followed by per oral antibiotic (levofloxacin and metronidazole) with only per oral antibiotics (moxifloxacin). Before randomization, the diagnosis of acute uncomplicated appendicitis is confirmed with a CT scan.

The hypothesis is that broad-spectrum intravenous antibiotics requiring additional hospital resources are not necessary for the treatment of uncomplicated acute appendicitis and that per oral mono therapy is non-inferior to the combination of intravenous and per oral antibiotic therapy.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of abdominal pain in emergency departments and appendectomy is the most common emergency abdominal surgery. The lifetime risk of acute appendicitis in males is 8.6% and 6.7% in females. In Finland according to Stakes data there were 6 377 appendectomies (3242 in males, 3135 in females, median age 35 years) performed in 2010. The total number of days in hospital care was 16 111 days and the mean length of hospital stay was three days.

Although acute appendicitis is the most common reason for surgical emergency department visit, its diagnosis still remains challenging. The clinical diagnosis has previously been based on patient history, physical examination and laboratory findings as well as the clinical surgical diagnosis. Several scoring systems have been created to aid in the diagnosis of acute appendicitis18-20, but the accuracy of clinical diagnosis without preoperative imaging is about 76 - 80 % for combined patient groups of males and females.

As acute appendicitis has historically been thought to always progress to perforation requiring emergency appendectomy, high negative appendectomy rates even up to 40 % in some patient populations have been previously accepted as good surgical practice. For the last two decades, the use of dedicated imaging in acute abdomen in general and also in acute appendicitis has led to improved diagnostic accuracy.

Based on large epidemiological studies, it is now known that complicated (perforated) and uncomplicated (non-perforated) appendicitis have followed different epidemiological trends. These unassociated epidemiologic trends suggest different pathophysiology for the two form of appendicitis. The differential diagnosis is essential as patients with an uncomplicated acute appendicitis may not require surgical intervention and might experience even spontaneous resolution without perforation. The majority (approximately 80 %) of acute appendicitis cases are of uncomplicated nature.

Complicated acute appendicitis defined as a finding of a perforation, appendicolith, abscess or a suspicion of a tumor, requires emergency appendectomy with the exception of cases with abscess as they are often managed conservatively.

Appendicolith is a calcified fecal concretion in the appendix resulting in internal luminal obstruction and it is the most common form of complicated acute appendicitis. In the first randomized study by Vons et al. comparing operative treatment and antibiotic therapy using CT as a diagnostic inclusion criterion, the presence of an appendicolith in preoperative CT scan was the only factor that significantly increased the risk of complicated appendicitis and it was also the only factor associated with the failure of antibiotic therapy for acute appendicitis. Indeed, if Vons et al had excluded the patients with an appendicolith from their analysis, no significant difference in the incidence of post-intervention peritonitis between the treatment groups would have been noticed in their study.

CT imaging is the primary imaging modality and the golden standard in the diagnosis of acute appendicitis as it establishes the diagnosis with almost perfect diagnostic accuracy. The advantages of CT imaging are high accuracy, availability, ease of performance and interpretation, and that it is rarely affected by bowel gas, severe abdominal pain or extreme body habitus. The main disadvantage of CT is exposure to radiation.

The increased use of preoperative CT imaging has been evaluated thoroughly by evaluating its impact on the negative appendectomy rate reducing the number of unnecessary appendectomies. In 2010, a mandatory imaging guideline for suspected acute appendicitis was implemented in the Netherlands. After implementation the negative appendectomy rate dropped significantly from 23 % to 6 % (p<0.001) reducing the surgical complication rate from 20% to 14 % and resulting in average cost-per-patient decrease by 594€.

The favorable diagnostic performance of CT imaging has encouraged optimization of the protocol to minimize exposure to radiation through the development of low-dose CT protocols. Low-dose protocols balance with as low as reasonably achievable-principle while maintaining diagnostic accuracy. However, low-dose protocols with intravenous contrast are still not implemented in routine clinical practice. These protocols require more advanced optimization and validation because of the wider need for contrast enhanced assessment. Kim et al showed that contrast enhanced low-dose CT (median radiation dose 116mmGy in dose-length product) was not inferior to standard-dose contrast enhanced CT (median radiation dose 521 mmGy), with negative appendectomy rates of 3.5% and 3.2% respectively and no statistical significance in appendiceal perforation rates or patients requiring additional imaging.

The investigators have performed a prospective observational study (OPTICAP trial, NCT02533869, Ethical committee of Turku University Hospital approval) in order to optimize a low-dose CT scan for both diagnosing acute appendicitis and to differentiate uncomplicated acute appendicitis from a complicated acute appendicitis. In this study, phantom imaging with 15 different imaging protocols were performed aiming to minimize radiation with optimal diagnostic accuracy. The phantom protocols were assessed by blinded evaluation of two gastrointestinal radiologists and the two best performing protocols were chosen for the clinical phase. The clinical evaluation included performing both of these imaging protocols for patients with suspected uncomplicated acute appendicitis evaluated by a senior digestive surgeon. All of the enrolled patients underwent laparoscopic appendectomy to evaluate the sensitivity and specificity of the imaging protocols. The most optimal imaging protocols were selected for use in the APPAC II trial; one low-dose CT protocol for patients with BMI under 30 and one optimised standard CT protocol for patients with BMI exceeding 30.

For over a century appendectomy has been the standard treatment for all patients with acute appendicitis. However, the results of our APPAC trial have now shown that the majority (73%) of patients with uncomplicated acute appendicitis were successfully treated with antibiotics alone. We also showed that none of the patients treated initially with antibiotics and later undergoing appendectomy had major complications or increased morbidity defining antibiotic therapy as a safe first-line treatment. Patients with a complicated acute appendicitis require emergency appendectomy and early identification of these patients is of vital importance. Laparoscopic appendectomy has become the golden standard for appendectomy providing lower morbidity and faster recovery compared with open appendectomy. For patients with uncomplicated acute appendicitis, the time has come to evaluate abandoning routine appendectomy and evaluating the optimal use of antibiotic therapy.

The aim of study is to optimize the antibiotic therapy for uncomplicated acute appendicitis by evaluating the success of treatment in both study groups and by comparing intravenous antibiotic therapy followed by per oral antibiotics with per oral antibiotic monotherapy. The study hypothesis is that broad-spectrum intravenous antibiotics requiring additional hospital resources are not necessary for the treatment of uncomplicated acute appendicitis and that per oral monotherapy is non-inferior to the combination of intravenous and per oral antibiotic therapy. The secondary aim is to evaluate the results of the randomized APPAC trial in a prospective patient cohort by implementing antibiotic therapy as the first-line treatment for uncomplicated acute appendicitis in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* CT confirmed uncomplicated acute appendicitis
* Ability to give consent to participate in the study

Exclusion Criteria:

* Age under 18 years or over 60 years
* Pregnancy or lactation
* Allergy to contrast media or iodine
* Allergy or contraindication to antibiotic therapy
* Renal insufficiency
* Metformin medication
* Severe systemic illness (for example malignancy, medical condition requiring immunosuppressant medication)
* CT confirmed complicated acute appendicitis
* Inability to co-operate and give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 552 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 1 year
  The resolution of acute uncomplicated appendicitis with allocated antibiotic treatment. Treatment success is defined as discharge from the hospital without the need for surgical intervention after the primary hospitalisation and no recurrent appendicitis during one-year follow-up.

SECONDARY OUTCOMES:
Late recurrence of appendicitis after antibiotic treatment | 1 year
  Recurring appendicitis after primary treatment considered successful, thus recurrence after one year
Duration of hospital stay | 1 month
  Hospital stay
Post-intervention complications | 10 years
  Complications according to the Clavien-Dindo classification
VAS pain score (visual analogue score) | 10 years
  Pain as described with a scale from 0-10
Sick leave | 1 month
  Duration of sick leave
Treatment costs | 1 year
  Treatment costs including hospital stay costs, medicinal costs, imaging costs, costs to treat possible complications, operative costs

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selanne L, Hurme S, Sippola S, Rautio T, Nordstrom P, Rantanen T, Pinta T, Ilves I, Mattila A, Savela EL, Rintala J, Paajanen H, Gronroos J, Haijanen J, Salminen P. Prognostic factors associated with primary non-responsiveness to antibiotics and appendicitis recurrence for CT-diagnosed uncomplicated acute appendicitis: secondary analysis of two randomized clinical trials. Br J Surg. 2025 Jul 3;112(7):znaf143. doi: 10.1093/bjs/znaf143. PMID 40741675
- [Derived] Selanne L, Haijanen J, Sippola S, Hurme S, Rautio T, Nordstrom P, Rantanen T, Pinta T, Ilves I, Mattila A, Rintala J, Marttila H, Merilainen S, Laukkarinen J, Savela EL, Paajanen H, Gronroos J, Salminen P. Three-Year Outcomes of Oral Antibiotics vs Intravenous and Oral Antibiotics for Uncomplicated Acute Appendicitis: A Secondary Analysis of the APPAC II Randomized Clinical Trial. JAMA Surg. 2024 Jul 1;159(7):727-735. doi: 10.1001/jamasurg.2023.5947. PMID 38630471
- [Derived] Sippola S, Haijanen J, Gronroos J, Rautio T, Nordstrom P, Rantanen T, Pinta T, Ilves I, Mattila A, Rintala J, Loyttyniemi E, Hurme S, Tammilehto V, Marttila H, Merilainen S, Laukkarinen J, Savela EL, Savolainen H, Sippola T, Aarnio M, Paajanen H, Salminen P. Effect of Oral Moxifloxacin vs Intravenous Ertapenem Plus Oral Levofloxacin for Treatment of Uncomplicated Acute Appendicitis: The APPAC II Randomized Clinical Trial. JAMA. 2021 Jan 26;325(4):353-362. doi: 10.1001/jama.2020.23525. PMID 33427870
- [Derived] Haijanen J, Sippola S, Gronroos J, Rautio T, Nordstrom P, Rantanen T, Aarnio M, Ilves I, Hurme S, Marttila H, Virtanen J, Mattila A, Paajanen H, Salminen P; APPAC study group. Optimising the antibiotic treatment of uncomplicated acute appendicitis: a protocol for a multicentre randomised clinical trial (APPAC II trial). BMC Surg. 2018 Dec 17;18(1):117. doi: 10.1186/s12893-018-0451-y. PMID 30558607